CLINICAL TRIAL: NCT05752825
Title: Acromegaly: Balance, Falls and Fracture Risk
Status: Completed | Type: Observational
Sponsor: Christian Alexander H Rosendal (Other)
Collaborators: Ipsen (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Christian Alexander H Rosendal, MD, PhD student at dept. of Endocrinology, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20220041
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acromegaly
Keywords: Joint disease; Bone disease; Fall risk; Fracture risk
MeSH Terms: conditions — Acromegaly; Joint Diseases; Bone Diseases | interventions — Absorptiometry, Photon; Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood samples will be stored in a research biobank for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acromegalic patients: Subjects with acromegaly
  Interventions: Radiation: HR-pQCT; Radiation: DXA scan; Diagnostic Test: Bone microindentation; Diagnostic Test: Hand grip and leg extension strength; Diagnostic Test: Timed up-and-go test; Diagnostic Test: Stabilometry; Diagnostic Test: Nerve conduction test; Diagnostic Test: Visual acuity test
- Healthy controls: Subjects without acromegaly
  Interventions: Radiation: HR-pQCT; Radiation: DXA scan; Diagnostic Test: Bone microindentation; Diagnostic Test: Hand grip and leg extension strength; Diagnostic Test: Timed up-and-go test; Diagnostic Test: Stabilometry; Diagnostic Test: Nerve conduction test; Diagnostic Test: Visual acuity test

INTERVENTIONS:
Radiation: HR-pQCT — HR-pQCT is a 3-dimensional imaging modality that can be applied to bone and joints in vivo, in order to non-invasively assess the quantity and quality of trabecular and cortical bone compartments separately. HR-pQCT will be applied to peripheral skeletal sites, namely the distal radius and tibia, where image slices equivalent to 9 mm of bone will be acquired. From this, parameters such as volumetric bone mineral density (vBMD), cortical density, cortical porosity, trabecular density, trabecular thickness, trabecular spacing and others will be calculated using specialized software. In the same scanning session, images of the wrist and ankle joints will be produced and analyzed for features of arthrosis, such as erosions, osteophytosis and others.
  Other Names: High Resolution peripheral Quantitative Computed Tomography
Radiation: DXA scan — Through DXA scans, we will obtain information regarding body composition, hip and spine bone mineral density, as well as examine any previous vertebral fractures using vertebral fracture assessment (VFA). VFA is a function of DXA scanners which allows for visualization of thoracic and lumbar vertebrae (usually T4-L4) in order to detect vertebral fractures34. Vertebral fractures can then be classified as either mild, moderate or severe using the method described by Genant et al35.
  Other Names: Dual X-ray Absorptiometry
Diagnostic Test: Bone microindentation — Using the OsteoProbe®, we will by microindentation measure the bone material strength index (BMSi), an in vivo surrogate measure of the fracture resistance of the cortical bone in the tibia. The participant is placed in a supine position with the examined leg rotated slightly outward. After identifying the site of interest, located midway between the medial tibial plateau and the medial malleolus, disinfectant is applied to the skin of the tibia being examined. Finally, under local anesthesia and fully sterile conditions, a test probe is inserted through the skin and onto the midshaft of the tibia, and the fracture resistance of the bone tissue is measured.
  Other Names: OsteoProbe
Diagnostic Test: Hand grip and leg extension strength — Hand grip strength will be assessed using a digital hand dynamometer as a measure of peripheral muscle strength. Leg extensor strength will be examined using the peak torque measured by an isometric dynamometer mounted on a fixed chair. 3 attempts will be given for each method, and the maximum value recorded.
Diagnostic Test: Timed up-and-go test — The TUG test is a functional test frequently used to assess balance in older individuals and is performed by measuring the time it takes for an individual to go from sitting to standing position, walk 3 meters, turn around and return to sitting position. A TUG score of >13,5 seconds is associated with an increased risk of falls.
Diagnostic Test: Stabilometry — Postural control will be assessed by means of a force platform that registers Center of Pressure (CoP) as a measure of postural stability. Measurements are performed under a variety of conditions, including eyes open/closed and on different surfaces. From the CoP measurements, parameters such as CoP range and CoP velocity in both antero-posterior and medial-lateral directions will be calculated using specialized software.
  Other Names: Balance board
Diagnostic Test: Nerve conduction test — To fully examine all components of balance, nerve conduction will be tested using a handheld device called NC-stat DPN-Check in order to assess any peripheral neuropathy.
Diagnostic Test: Visual acuity test — Visual acuity will be tested using an automated refractometer (KR-800S Auto-kerato-refractometer, Topcon Healthcare, The Netherlands).

SUMMARY:
The goal of this observational, cross-sectional study is to study bone quality, joint quality and fall risk in acromegalic patients, compared with healthy controls. The main questions it aims to answer are:

* what is the optimal method for evaluating bone quality and fracture risk in acromegalic patients?
* are acromegalic patients at increased risk of falling?
* is HR-pQCT a feasible method for evaluating acromegalic joint disease? Participants will undergo HR-pQCT scans, DXA scans, OsteoProbe examination and fall risk assessments. Results will be compared to matched healthy controls.

DETAILED DESCRIPTION:
Patients with an established diagnosis of acromegaly will be recruited from March 2023 to March 2025. Patients will be informed of the study during scheduled visits to the pituitary endocrinology outpatient clinic at Aalborg University Hospital by one of two specialists in pituitary endocrinology. Patients will be given information regarding the study, and if interested, they will be provided with a form to fill out with their contact information, so they can be contacted by the investigators or other staff affiliated with the study. Should the patient agree to be contacted via telephone or e-mail, they will be given an instruction regarding their rights as a participant in a scientific study ("Dine rettigheder som forsøgsperson i et sundhedsvidenskabeligt forskningsprojekt") as well as written material specifically pertaining to the study ("Deltagerinformation"). Should the subject be deemed fit for the study, based on the in- and exclusion criteria, contact will be made via phone or e-mail and they will receive further information regarding the study, and offered a personal meeting with one of the investigators, where details of the study procedures will be outlined. The meeting will take place in a dedicated, undisturbed office at the disposition of the Department of Endocrinology, in order to ensure due privacy during the meeting. In advance, the subject will be informed of the opportunity to bring a relative or other representative to the meeting. At the meeting, the participant and any representative will be informed of the 24-hour deliberation period before providing informed consent. No study procedures will be performed until the informed consent form has been signed by both the participant and the investigator.

As mentioned above, healthy controls will be recruited via the aforementioned database, social media and websites such as www.forsoegsperson.dk. Potential participants who contact the principal investigator through these channels will be provided with written material pertaining to the study ("Deltagerinformation") and a description of their legal rights as a participant ("Dine rettigheder som forsøgsperson i et sundhedsvidenskabeligt forskningsprojekt"). Should the potential participant meet the in- and exclusion criteria, they will be invited to a personal meeting, where details of the study are explained, having been informed of the opportunity to bring a representative or relative to the meeting in advance. Should they wish to participate, a 24-hour deliberation period will be given prior to obtaining written informed consent.

After providing informed consent, the participants will undergo a series of study procedures. Bone quality will be assessed by way of High-Resolution peripheral Quantitative Computed Tomography (HR-pQCT) images of the distal radius and tibia. Bone material strength index (BMSi) is assessed using an OsteoProbe. In addition to this, postural control will be assessed using a balance board to obtain a surrogate measure of fall risk. Body composition, bone mineral density and vertebral fracture assessment (VFA) will be analyzed via Dual X-ray Absorptiometry (DXA) scans and peripheral muscle strength will be assessed via hand grip strength and knee extension torque measurements, and visual acuity tested with standard methods. Data will be analyzed using relevant statistical analyses and presented as a cross-sectional study.

HIGH RESOLUTION PERIPHERAL QUANTITATIVE COMPUTED TOMOGRAPHY (HR-PQCT) HR-pQCT is a 3-dimensional imaging modality that can be applied to bone and joints in vivo, in order to non-invasively assess the quantity and quality of trabecular and cortical bone compartments separately. HR-pQCT will be applied to peripheral skeletal sites, namely the distal radius and tibia, where image slices equivalent to 9 mm of bone will be acquired. From this, parameters such as volumetric bone mineral density (vBMD), cortical density, cortical porosity, trabecular density, trabecular thickness, trabecular spacing and others will be calculated using specialized software. In the same scanning session, images of the wrist and ankle joints will be produced and analyzed for features of arthrosis, such as erosions, osteophytosis and others.

The scanner's gantry is relatively narrow and shallow (rear physical stop) only allowing the distal peripheral skeleton to be accommodated. The limb being scanned is immobilized in a carbon fiber shell. A scout view, essentially a two-dimensional x-ray scan, is obtained so that the operator can identify a precise region for the three-dimensional measurement. Because HR-pQCT uses a polychromatic X-ray source it is subject to beam hardening as well as scatter artefacts, which can significantly impact geometric and densitometric measures. Once the images have been acquired, a default patient evaluation protocol is used to analyze the scans over the entire 9 mm three-dimensional region to assess a wide range of standard and optional structural and density parameters.

The effective radiation dose for one HR-pQCT scan at the distal tibia or radius is 0,003 - 0,005 mSv, which is considered a low radiation dose33. In comparison, a regular chest X-ray yields a dose of 0,01 - 0,1 mSv and dental X-ray yields 0,005 mSv. The worldwide average effective radiation dose from natural background radiation is 2,4 mSv per year. The average effective radiation dose in Denmark is 3 mSv per year.

Estimated time: 30 min. WHOLE BODY DUAL X-RAY ABSORPTIOMETRY (DXA) SCAN AND VERTEBRAL FRACTURE ASSESSMENT Through DXA scans, we will obtain information regarding body composition, hip and spine bone mineral density, as well as examine any previous vertebral fractures using vertebral fracture assessment (VFA). VFA is a function of DXA scanners which allows for visualization of thoracic and lumbar vertebrae (usually T4-L4) in order to detect vertebral fractures34. Vertebral fractures can then be classified as either mild, moderate or severe using the method described by Genant et al35.

The effective radiation dose is between 0,001 and 0,01 mSv for one whole body DXA scan, between 0,003 and 0,03 mSv for one hip and lumbar spine DXA scan and 0,003 mSv for one VFA scan. As such, the total effective radiation dose for the DXA scans is between 0,007 and 0,043 mSv.

The whole body DXA scan, hip and lumbar spine DXA scan and VFA scan will be performed consecutively.

Estimated time: 50 min. MICROINDENTATION, BONE MATERIAL STRENGTH INDEX (BMSI) AND THE OSTEOPROBE® Using the OsteoProbe®, we will by microindentation measure the bone material strength index (BMSi), an in vivo surrogate measure of the fracture resistance of the cortical bone in the tibia. The participant is placed in a supine position with the examined leg rotated slightly outward. After identifying the site of interest, located midway between the medial tibial plateau and the medial malleolus, disinfectant is applied to the skin of the tibia being examined. Finally, under local anesthesia and fully sterile conditions, a test probe is inserted through the skin and onto the midshaft of the tibia, and the fracture resistance of the bone tissue is measured. Without removing the probe from the skin, this process is repeated a minimum of eight (maximally 18) times to provide a sufficient number of measurements. By means of a synthetic polymer calibration phantom, the BMSi is calculated via specialized software provided by the manufacturer. After the procedure, a sterile bandage will be applied to the puncture site and all sharp and/or biohazardous materials will be disposed of in an appropriate manner.

Estimated time: 20 min. HAND GRIP STRENGTH (HGS) AND LEG EXTENSION STRENGTH Hand grip strength will be assessed using a digital hand dynamometer as a measure of peripheral muscle strength. Leg extensor strength will be examined using the peak torque measured by an isometric dynamometer mounted on a fixed chair. 3 attempts will be given for each method, and the maximum value recorded.

Estimated time: 10 min. TIMED UP-AND-GO (TUG) The TUG test is a functional test frequently used to assess balance in older individuals and is performed by measuring the time it takes for an individual to go from sitting to standing position, walk 3 meters, turn around and return to sitting position. A TUG score of >13,5 seconds is associated with an increased risk of falls.

Estimated time: 10 min. STABILOMETRY Postural control will be assessed by means of a force platform that registers Center of Pressure (CoP) as a measure of postural stability. Measurements are performed under a variety of conditions, including eyes open/closed and on different surfaces. From the CoP measurements, parameters such as CoP range and CoP velocity in both antero-posterior and medial-lateral directions will be calculated using specialized software.

Estimated time: 20 min. NERVE CONDUCTION TEST To fully examine all components of balance, nerve conduction will be tested using a handheld device called NC-stat DPN-Check in order to assess any peripheral neuropathy.

Estimated time: 10 min. VISUAL ACUITY TEST Visual acuity will be tested using an automated refractometer (KR-800S Auto-kerato-refractometer, Topcon Healthcare, The Netherlands).

Estimated time: 10 min. Our laboratory has ample experience and know-how regarding the above-mentioned methods and their application in different patient groups.

QUESTIONNAIRES Through questionnaires we will obtain information regarding previous falls and fractures, overall quality of life (Acro-QoL), joint-related symptoms (Western Ontario and McMaster universities osteoarthritis Index, WOMAC), fear of falling (Falls Efficacy Scale International, FES-I) and balance (Berg Balance Scale). Medicine lists will be collected from all participants.

BIOCHEMICAL BONE MARKERS AND BLOOD SAMPLES To assess biochemical markers of bone metabolism, we will measure fasting serum levels of procollagen-1 N-terminal propeptide (P1NP, a marker of bone formation) and cross-linked C telopeptide of type I collagen (CTX, a marker of bone resorption) as well as sclerostin (an inhibitor of bone formation). To assess other hormones with influence on bone quality, we will measure levels of vitamin D and parathyroid hormone (PTH). In total, a volume of approximately 16mL of blood (4x 4mL vials) will be collected from each participant, both acromegalic and controls. For practical reasons, these blood samples are frozen after collection, stored in a research biobank, and analyzed in one session upon all participants' completion of the study procedures. Before analysis, Danish Tissue Utilization Register (Vævsanvendelsesregistret) will be consulted; should the participant be listed herein, the blood sample will not be analyzed. After analysis, any remaining material will be destroyed.

Two extra vials of blood (10mL total) will be extracted and stored in a biobank for future research, to enable analysis of any future bone markers or other biomarkers of interest for this project. An application will be submitted to the Danish Data Protection Agency in this regard. Blood samples will be frozen and stored in an encrypted fashion and in compliance with the Danish Data Protection Act for 15 years after completion of the study, or until their destruction is requested by the participant. Blood samples will be collected from both acromegalic subjects and healthy controls, in order to determine differences in biochemical markers between acromegalic subjects and control subjects. Participants will be asked to sign a separate consent form regarding storage of their biological material (blood sample) in a biobank for future research.

All blood samples are stored in a freezer at -80 degrees Celsius.

ELIGIBILITY:
Inclusion Criteria:

1. Verified acromegaly diagnosis
2. Age >18 years
3. Ability to provide informed consent
4. Ability to stand on both legs for >5 minutes at a time and walk >6 meters
5. Patient is eugonadal, either naturally or by hormone replacement therapy

Exclusion Criteria:

1. Established diagnosis of severe kidney or liver dysfunction, malabsorption, multiple myeloma or other diseases associated with reduced bone quality
2. Treatment with supraphysiological doses of glucocorticoids or other drugs that impair bone quality
3. Diagnosis of rheumatoid arthritis, psoriatic arthritis or other joint diseases unrelated to acromegaly
4. Active drug or alcohol abuse
5. Pregnancy
6. Known allergy/hypersensitivity to local anaesthetics or disinfectant
7. Other factors that render the subject unable to participate in the clinical study, based on the judgment of the investigator(s)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acromegaly who attend the Neuroendocrinology outpatient clinic at Aalborg University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Bone material strength index | 20 min
  Measured by micro indentation
Volumetric BMD | 30 min
  Measured by HR-pQCT
Area BMD | 50 min
  Measured by DXA

SECONDARY OUTCOMES:
Balance (center of pressure and sway) | 20 min
  Measured by force platform
Visual acuity | 15 min
  Measured by auto-kerato-refractometer
Nerve conduction velocity | 5 min
  Measured by handheld device
Muscle strength | 10 min.
  Hand grip and leg extension, Measured by dynamometers

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be made available upon request after the study has concluded.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT05752825/Prot_SAP_000.pdf